CLINICAL TRIAL: NCT00345670
Title: A Phase I, Randomized, Double-Blind, Placebo-Controlled, Dose-Escalation Study to Evaluate the Safety, Tolerability, Immunogenicity, and Viral Shedding of MEDI-534, a Live, Attenuated Intranasal Vaccine Against Respiratory Syncytial Virus (RSV) and Parainfluenza Virus Type 3 (PIV3), in Healthy RSV and PIV3 Seropositive 1-9 Year-Old Children
Brief Title: Study to Evaluate the Safety of MEDI-534 Vaccine Against Respiratory Syncytial Virus (RSV) and Parainfluenza Virus Type 3 (PIV3) in Healthy Children
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: MedImmune LLC (Industry)
Responsible Party: Margarita M Gomez, M.D., MedImmune LLC
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: MI-CP130
Record Dates: First submitted 2006-06-27; First posted 2006-06-28 (Estimated); Last update posted 2008-09-03 (Estimated); Status verified 2008-09

CONDITIONS: Healthy
Keywords: Lower respiratory tract illness; RSV and PIV3 infection

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- 1 (Experimental): MEDI-534
  Interventions: Biological: MEDI-534
- 2 (Experimental): MEDI-534
  Interventions: Biological: MEDI-534
- 3 (Experimental): MEDI-534
  Interventions: Biological: MEDI-534

INTERVENTIONS:
Biological: MEDI-534 — 10:4 TCID50 of MEDI-534 intranasal spray Study Day 0
  Arms: 1
Biological: MEDI-534 — 10:5 TCID50 of MEDI-534 intranasal spray Study Day 0
  Arms: 2
Biological: MEDI-534 — 10:6 TCID50 of MEDI-534; intranasal spray
  Arms: 3

SUMMARY:
This is a randomized, double-blind, placebo-controlled, dose-escalation, Phase 1, multi-center study to evaluate the safety, tolerability, immunogenicity, and viral shedding of MEDI-534 in healthy children 1-9 years of age who are seropositive for respiratory syncytial virus (RSV) and parainfluenza virus type 3 (PIV3) at screening.

DETAILED DESCRIPTION:
This is a randomized, double-blind, placebo-controlled, dose-escalation Phase 1 multi-center study to evaluate the safety, tolerability, immunogenicity, and viral shedding of MEDI-534 in healthy children 1-9 years of age who are seropositive for RSV and PIV3 at screening. MEDI-534 will be administered at dosage levels of 10:4 TCID50, 10:5 TCID50, or 10:6 TCID50 to three cohorts of subjects in a staggered, step-wise fashion. A single dose of study vaccine (MEDI-534 or matched volume of vehicle placebo) will be administered on Study Day 0 by nasal spray, one-half dose into each nostril. The target sample size is 120 subjects randomized 1:1 (MEDI-534 to placebo), with 40 subjects in each of three cohorts. Randomization will be stratified by site. This study will enroll during the RSV off season at multiple sites in the United States and Chile.

ELIGIBILITY:
Inclusion Criteria:

* Male or female aged 1 through 9 years old
* In general good health
* Seropositive for RSV (enzyme-linked immunosorbent assay [ELISA] titer > 12 U/ml) and PIV3 (hemagglutination-inhibition [HAI] titer > 1:8)
* Subject's parent/legal representative available by telephone
* Written informed consent and Health Insurance Portability and Accountability Act (HIPAA) authorization (if applicable) obtained from the subject's parent/legal representative
* Ability of the subject's parent/legal representative to understand and comply with the requirements of the protocol as judged by the investigator
* Ability to complete the follow-up period of 6 months following dosing as required by the protocol

Exclusion Criteria:

* Any fever and/or respiratory illness (e.g., cough or sore throat) within 7 days prior to randomization
* Any drug therapy (chronic or other) within 7 days prior to randomization or expected receipt of such therapy through the protocol-specified blood collection 28-35 days after study vaccine dosing
* Any current or expected receipt of systemic immunosuppressive agents including steroids; children in this category should not receive study vaccine until immunosuppressive agents including corticosteroid therapy have been discontinued for less than or equal to 30 days
* Receipt of blood transfusion within 7 months prior to randomization or expected receipt through 35 days after study vaccine dosing
* Receipt of immunoglobulin products within 11 months prior to randomization or expected receipt through 35 days after study vaccine dosing
* Receipt of any investigational drug within 60 days prior to randomization or expected receipt through 180 days after study vaccine dosing
* Receipt of any other live virus vaccine within 30 days prior to randomization or expected receipt through the protocol-specified blood collection 28-35 days after study vaccine dosing
* Receipt of any inactivated (i.e., non-live) vaccine within 14 days prior to randomization or expected receipt through the protocol-specified blood collection 28-35 days after study vaccine dosing
* History of Guillain-Barré syndrome
* Known or suspected immunodeficiency, including HIV
* Known or suspected acute or chronic hepatitis infection
* Living at home or attending day care with children less than or equal to 24 months of age
* Contact with pregnant caregiver
* Household contact who is immunocompromised; the subject should also avoid close contact with immunocompromised individuals for at least 30 days after study vaccine dosing
* History of hypersensitivity to kanamycin or other aminoglycoside antibiotics (gentamicin, tobramycin, etc)
* Previous medical history, or evidence, of chronic illness may compromise the safety of the subject
* At screening any of the following laboratory tests outside of the laboratory normal range: complete blood count (CBC) with differential and platelet count, AST, ALT, blood urea nitrogen (BUN), creatinine, or other abnormal laboratory value in the screening panel that, in the opinion of the principal investigator, is considered to be clinically significant or may potentially compromise the safety of the subject during the conduct of the study
* History of medically confirmed diagnosis of asthma, reactive airway disease, or chronic obstructive pulmonary disease (COPD)
* Passive primary household smoking
* Family member or household contact who is an employee of the research center with the conduct of the study
* Any condition that, in the opinion of the investigator, might interfere with study vaccine evaluation

Ages: 1 Year to 9 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 120
Dates: Start 2006-06; Study Completion 2007-05 (Actual)

PRIMARY OUTCOMES:
To describe the safety and tolerability of 1-9 year old RSV and PIV3 seropositive children | Day 28
Reactogenicity evaluations (REs) from administration of study vaccine through 28 days post-dosing | Day 28 post final vaccination
Adverse events (AEs) from administration of study vaccine through 28 post-dosing | Day 28 post final vaccination
Serious adverse events (SAEs) from administration of study vaccine through 28 days post-dosing | Day 180

SECONDARY OUTCOMES:
To describe the immunogenicity and viral shedding of MEDI-534 | Days 3, 7, 14 days (± 1 day) and 28 35 days after study vaccine dosing as well as at any unscheduled study visits.
The viral shedding of MEDI-534 will be assessed by the absence or presence of vaccine-type virus from nasal swab and nasal wash samples | Days 3, 7, 14 days (± 1 day) and 28 35 days after study vaccine dosing as well as at any unscheduled study visits.

CONTACTS AND LOCATIONS:
Overall Officials: Margarita M Gomez, M.D., Study Director — MedImmune LLC
Locations (12):
- United States (12):
  - Edinger Medical Group, Fountain Valley, California
  - Heart of America Research, Shawnee, Kansas
  - Heart of America Research, Topeka, Kansas
  - Kentucky Pediatric/Adult Research, Bardstown, Kentucky
  - Cincinnati Children's Hospital Medical Center, Division of Infectious Disease, Crestview Hills, Kentucky
  - University of Maryland Pediatric Ambulatory Center, Baltimore, Maryland
  - Meridian Clinical Research, LLC, Omaha, Nebraska
  - Regional Clinical Research, Inc., Binghamton, New York
  - Children's Hospital at Montefiore; Montefiore Medical Center, The Bronx, New York
  - Pediatric Associates of Mt. Carmel, Inc., Cincinnati, Ohio
  - Primary Physicians Research, Inc., Pittsburgh, Pennsylvania
  - University Physicians Internal Medicine, Huntington, West Virginia

REFERENCES:
- [Derived] Gomez M, Mufson MA, Dubovsky F, Knightly C, Zeng W, Losonsky G. Phase-I study MEDI-534, of a live, attenuated intranasal vaccine against respiratory syncytial virus and parainfluenza-3 virus in seropositive children. Pediatr Infect Dis J. 2009 Jul;28(7):655-8. doi: 10.1097/INF.0b013e318199c3b1. PMID 19483659